CLINICAL TRIAL: NCT06438029
Title: The Effect of Education Given to Nursing Students on Their Perceptions of Disaster Response Competence: A Randomized Controlled Trial
Brief Title: The Effect of Disaster Training on the Perception of Disaster Response Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FATOŞ UNCU (Other)
Responsible Party: Sponsor-Investigator, FATOŞ UNCU, assistant professor, Firat University
Organization: Firat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FU-SBF-FU-02
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Public Health Nursing
Keywords: Natural disasters; Nursing students
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This research is a randomised control study with pretest-posttest design.
Who Masked: Participant, Investigator
Masking Description: Randomisation method will be used to determine how the experimental and control groups will be separated at the beginning of the study (13). As the randomisation method, "simple randomisation method" was chosen in order to provide equal number of samples in two groups. Randomisation will be performed using https://www.randomizer.org/ website in computer environment. According to the randomisation outputs, the individuals to be included in the experimental and control groups will be listed. Columns between 1-90 will be created in the system. Patients will be randomly assigned to the groups by considering the numbers 1 and 2 in the columns (nursing education group 1 and control group 2).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): The forms used in the study were collected by the researcher through face-to-face interviews in seminar halls in schools. Firstly, the students in the experimental group will be trained on disaster and disaster response. The trainings were organised as a total of four sessions with a two-week interval of twenty minutes in each session. Personal Information Form and Disaster Intervention Self-Efficacy Scale were filled as pre-test in the seminar halls of the schools under the supervision of the researcher.
  Interventions: Other: Education group; Other: control group
- Control group (No Intervention): Personal Information Form and Disaster Response Self-Efficacy Scale will be applied to the students in the control group as a pre-test. No training will be given to the control group. In the last stage of the research, the Disaster Response Self-Efficacy Scale will be applied to the control group as a post-test and the data collection process will be terminated. After the last test was applied to the groups, training materials will be given to the people who demanded from the control group.

INTERVENTIONS:
Other: Education group — the students in the experimental group will be trained on disaster and disaster response
  Arms: Education group
Other: control group — the students in the experimental group will be trained on disaster and disaster response
  Arms: Education group

SUMMARY:
Due to the increase in disasters, humanity is facing an increasing threat to life and property. Disasters occur with little warning and can last for hours or months. Existing literature reveals that most nurses are not prepared for a disaster in the community. Continuous preparedness requires the involvement of staff and nursing students in the development, review and implementation of the disaster plan. The development of ongoing, easily accessible, engaging and realistic educational programmes is best for the acquisition of skills and competence. An experimental study with pretest-posttest control group The project is planned to be conducted with the fourth grade students of the Department of Nursing, Faculty of Health Sciences, Fırat University in a randomised controlled study model with pre-test-post-test control group. The population of the study will consist of the fourth year students of the Department of Nursing, Faculty of Health Sciences, Fırat University. The sample will consist of 90 students with 0.05 error, 0.95 confidence interval, 0.95 confidence interval, 0.6 effect size and 0.80 representation power of the universe with the power analysis. These students will be divided into 45 experimental and 45 control groups. In the first stage of the study, the experimental and control group students were asked to complete the "Personal Information Form" and '' Disaster response self-efficacy scale" will be filled. In the second stage of the research, the students in the experimental group will be given a detailed and planned training programme. After the training, the students

DETAILED DESCRIPTION:
Natural disasters, which cause a large number of casualties, increase the workload and lead to disability of individuals, have always been an important public health problem. Natural disasters are unpredictable and often sudden events that cause great destruction and loss of life and severe psychological symptoms for survivors. Disaster preparedness refers to all previous action plans and efforts to establish a disaster response system before a disaster occurs. To be prepared, nurses need to have sufficient knowledge and skills to minimise the negative effects of a disaster, including trauma, infectious diseases, physical and psychological distress. However, there is evidence that most nurses do not feel adequately prepared for a disaster in the community. In a study in which the general knowledge levels of nurses in developing countries about disaster preparedness were evaluated, the knowledge and skills of nurses especially in the Asia-Pacific Region about disasters were found to be inadequate. In another study, it was reported that Iranian nurses had inadequate knowledge about disaster preparedness.

Despite the increasing number of disasters all over the world and the warnings of international nursing organisations and the World Health Organisation about the preparedness of nurses for disasters, it is seen that the training of nurses for disasters is inadequate and studies on this subject are limited.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th year Nursing Student
* Want to participate in the research voluntarily

Exclusion Criteria:

* Student wants to leave the study
* Incomplete filling of survey forms

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Disaster response self-efficacy scale: | 3 month
  The scale is a 5-point Likert type and consists of a total of 19 items and 3 sub-dimensions (On-site rescue competence, Disaster psychological nursing competence, Nature of the role undertaken in disaster and adaptation competence). The scale is answered as having no self-confidence (1 point), basically no self-confidence (2 points), some self-confidence (3 points), basically self-confident (4 points) and full self-confidence (5 points). The scale score is calculated by summing the answers to the questions. A high score from the scale indicates high disaster response self-efficacy. In the Turkish validity and reliability study of the scale, the Cronbach alpha coefficient was found to be 0.96.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)